CLINICAL TRIAL: NCT05000333
Title: The Consequences of Covid-19 on the Psychological and Physical Health of the Nursing Staff of the Hospital of Villeneuve Saint Georges and on Their Professional Activity. (SST-Covid Impact)
Brief Title: Consequences of Covid-19 on the Psychological and Physical Health of the Nursing Staff and on Their Professional Activity.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: SST-Covid Impact
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Work-related Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-questionnaire — The study will be proposed to caregivers who work at Centre Hospitalier Intercommunal de Villeneuve-Saint-Georges, who agree to answer the questionnaire anonymously

SUMMARY:
The aim of this research is to identify the consequences of the Covid-19 on the physical and psychological health of the nursing staff of the Intercommunal Hospital of Villeneuve-Saint-Georges and on their professional activity thanks to a self-questionnaire.

This anonymous self-questionnaire is intended for all the CHIV care workers who were infected by the coronavirus during the first wave and identified by the occupational health service.

DETAILED DESCRIPTION:
The covid-19 pandemic has had an important impact in the world, in France, it has put our health system under tension. We know that a health crisis of this magnitude can induce psychological and physical disorders, particularly in exposed caregivers.

Systematic occupational medicine consultations of all medical and paramedical personnel, whether tenured or not, working at the Villeneuve Saint Georges Hospital (CHIV) who presented a Covid-19 between February 1 and June 30, 2020, allowed us to note the presence of multiple after-effects.

The present study evaluates the consequences of the disease on the physical and psychological health of these caregivers and on their professional activity.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient
2. Part of the medical and paramedical staff working at the CHIV,
3. Having been reached by Covid-19 during the first wave, between February 1st and June 30th 2020.
4. Patient affiliated to a social security system

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care population (medical and paramedical) practicing at the Centre Hospitalier Intercommunal de Villeneuve-Saint-Georges, having been reached by the Covid-19 during the first wave, between February 1st and June 30th 2020.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Physical and psychological health | up to 1 month
  Percentage of physical and psychological after-effects

SECONDARY OUTCOMES:
Recognized occupational diseases | up to 1 month
  Number of recognized occupational diseases
Days of sick leave | up to 1 month
  Evaluate the number of days of sick leave.
Reclassifications | up to 1 month
  Evaluate the number of reclassifications
workstation adjustments | up to 1 month
  Evaluate the number workstation adjustments
Repercussions on the professional activity | up to 1 month
  The existence of repercussions on the professional activity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Villeneuve-Saint-Georges, Villeneuve-Saint-Georges, IDF, France

IPD SHARING:
Plan to Share IPD: No